CLINICAL TRIAL: NCT04952207
Title: Effectiveness and Safety of Direct-Acting Antiviral Agents for the Treatment of Chronic Hepatitis C: Multi-center, Prospective, Observational Real-world Study in EASTERN China
Brief Title: Effectiveness and Safety of Direct-Acting Antiviral Agents for the Treatment of Chronic Hepatitis C
Acronym: C-DIAMOND
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Qing XIe (Other)
Collaborators: Gilead Sciences (Industry); Tigermed Consulting Co., Ltd (Industry)
Responsible Party: Sponsor-Investigator, Qing XIe, Director of Department of Infectious Disease, Rui Jin Hospital, Ruijin Hospital
Organization: Ruijin Hospital (Other)
Other Study IDs: IN-CN-342-5424
Record Dates: First submitted 2021-06-24; First posted 2021-07-07 (Actual); Last update posted 2021-07-07 (Actual); Status verified 2021-07

CONDITIONS: Hepatitis C, Chronic
Keywords: Chronic hepatitis C; Direct-acting antiviral agents; Sustained virological response
MeSH Terms: conditions — Hepatitis C, Chronic | interventions — daclatasvir; asunaprevir; ombitasvir; paritaprevir; dasabuvir; Sofosbuvir; velpatasvir; ledipasvir; elbasvir; grazoprevir; danoprevir; glecaprevir; pibrentasvir; voxilaprevir

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 24 Weeks
Biospecimen Retention: Samples Without DNA — serum, HCV RNA
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- DAA Group: Chronic hepatitis C patients treated with DAA
  Interventions: Drug: Direct-acting antiviral agents

INTERVENTIONS:
Drug: Direct-acting antiviral agents — The initial DAA treatment and its dose for all patients is determined by the infectionist or hepatologist based on the clinical diagnosis and treatment routine. The administration dose in the instructions for use for current DAAs marketed in China Mainland unnecessary to combine with any IFN is shown but not limited as follows: Sofosbuvir, Ombitasvir/Paritaprevir/Ritonavir, Dasabuvir, Daclatasvir, Asunaprevir, Elbasvir/Grazoprevir, Sofosbuvir/Velpatasvir and Ledipasvir/Sofosbuvir.
  Other Names: daclatasvir; asunaprevir; ombitasvir; paritaprevir; dasabuvir; sofosbuvir; velpatasvir; ledipasvir; elbasvir; grazoprevir; danoprevir; glecaprevir; pibrentasvir; voxilaprevir

SUMMARY:
Clinical trials evaluating DAA have shown excellent rates of SVR and good safety profiles in patients with CHC infection. Real world data from TARGET, TRIO, IFI, DHCR, DALTON-C, as well as those cohorts from Japan, Taiwan and Korea further confirmed clinical trial findings of DAA in routine practice where populations are more complex. However, these populations are different from Chinese for different host and virus characteristics which limit the applicability of results to local practice.

As DAA launched in China since 2017, the availability of INF free DAA treatment will likely lead to better treatment outcome in routine practice, but there are currently no data available to test the hypothesis.

In clinical practice, the uptake of DAA regimen will depend on a combination of physician preference, patient's characteristics and drug access. This study will also identify how these three variables affect DAA regimen uptake.

This study to 1) characterize pts receiving IFN free DAA regimens, 2) represent common practice in China, 3) describe outcome of various INF free DAA therapy, and 4) confirm registration study results.

DETAILED DESCRIPTION:
Chronic Hepatitis C (hereinafter referred to as "CHC") is a viral hepatitis caused by the infection of Hepatitis C virus (HCV). In 2007, a cross-sectional study in six cities showed that the prevalence of HCV was 0.58% in China. It was estimated that there were about 10 million HCV patients in our country. If hepatitis C was not treated in time, about 75% of patients would progress into chronic hepatitis C six months after virus infection; the probability was 5%~15% for progression into cirrhosis and 2%~4% for progression into hepatocellular carcinoma 20 years after the infection of chronic hepatitis C. One analysis of cirrhosis etiology in northern China found that the proportion of CHC-induced cirrhosis was increased from 6.39% in 2002 to 13.91% in 2011.

As a result of the severely epidemiological burden of CHC, the World Health Organization (WHO) has established a target to eliminate the hepatitis harm in 2030 ("2030 global targets" for short) that 90% reduction in new cases of chronic hepatitis B and C in 2030, 80% of treatment-eligible people with chronic hepatitis B and C treated and 65% reduction in hepatitis B and C deaths. As a part of the strategy to achieve this target, WHO includes the treatment with direct-acting antiviral agents (DAAs) into the 2017 Essential Medicine List. In addition, the Viral Hepatitis Prevention and Control Programs in China (2017-2020) also emphasize the application of more effective treatment as a part of the strategy to reduce the transmission of HCV.

Direct-acting antiviral agents (DAAs) are a new drug for the treatment of CHC now. In 2017, China Food and Drug Administration (CFDA)/ National Medical Products Administration (NMPA) approved the marketing of Sofosbuvir of Gilead, Ombitasvir/Paritaprevir/Ritonavir Tablets + Dasabuvir of AbbVie, Daclatasvir Tablets + Asunaprevir Capsules of Bristol-Myers Squibb; Elbasvir/Grazoprevir of MSD, Sofosbuvir/Velpatasvir and Ledipasvir/Sofosbuvir of Gilead and Danoprevir of Ascletis in 2018. Before the DAAs are marketed, the pegylated interferon combined with ribavirin (PR) therapy is the major therapy of antiviral for HCV-infected patients. However, the real-world study showed that the sustained virological response (SVR) of PR therapy was 71.1%. The DAAs therapy was demonstrated with shorter treatment time, better efficacy, fewer adverse events, and higher compliance compared with the PR therapy.

Multiple clinical trials indicated a high SVR rate and safety of DAAs in CHC patients. The real-world studies with more complicated patient populations, including TARGET, TRIO, IFI, DHCR, and DALTON-C as well as the cohort studies from Japan, Taiwan, and the Republic of Korea also further demonstrated good clinical efficacy with DAAs. While GT 1-3 is prevalent worldwide, subtypes of 1b, 2a, 3a, 3b, and 6a are prevalent in China, and among them, GT 3 and 6 are expanding. Since the host and virus characteristics of these populations are different from the Chinese population, the BMI of the Chinese population is smaller than that of the European and American population, IL28 CC GT is predominant, and HCV patients of GT 3b is most common among HCV patients of GT 3. So, it is necessary to further demonstrate the applicability of the results of these studies to Chinese patients.

DAAs have been marketed in China since 2017. The treatment with DAAs unnecessary to combine with any interferon (IFN) may obtain better therapeutic effect in clinical practice. However, there is a lack of real-world data to verify this hypothesis now.

In clinical practice, the selection of therapy with DAAs will depend on the physician preference, patient baseline characteristics, and drug accessibility. This study will also determine the baseline status of patients receiving different DAA treatments and possible reasons for doctors' prescriptions in the real world.

In the eastern part of China, the GTs of HCV infected patients are GT 1b (69.2%), GT 2a (20.8%), GT 3a (2.2%), GT 3b (4.4%) and GT 6 (3.2%).To demonstrate whether DAAs provide good efficacy and safety to the patients, including the patients with cirrhosis, accompanying with infection, kidney/liver transplantation, or no response to PR therapy, the purpose of this study is to 1) describe the patient characteristics for DAA therapy unnecessary to combine with any IFN in routine clinical practice in China; 2) describe the therapeutic effect of multiple DAAs unnecessary to combine with any IFN to verify above hypothesis.

ELIGIBILITY:
Inclusion Criteria:

* All Chronic hepatitis C patients to be treated with the DAAs approved by CFDA/NMPA
* Age≥18 years

Exclusion Criteria:

* Patients experienced with DAAs
* Documented HCC, AFP>500ng/ml
* Unlikely to survive 1 year or inability to participate and follow up for the study period

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The primary objective of this study is to obtain the SVR12 rate of CHC patients in Eastern China. The previous study of Rui Jin Hospital Affiliated to Shanghai Jiao Tong University School of Medicine showed that the SVR12 rate was 0.988 (CI 95%: 0.952-1.0, Shanghai, China, Rui Jin Hospital, 26th APASL annual meeting, PO241). In this study, the estimated value of SVR is set to 95%, the bilateral significance level is 0.05 and the sampling error is 0.03. The estimated sample size is 225 as per the sample size calculation formula. Considering the patient withdrawal, this study is planned to collect 300 patients.
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2019-03-06 (Actual); Primary Completion 2021-07-31 (Estimated); Study Completion 2021-08-31 (Estimated)

PRIMARY OUTCOMES:
SVR12 rate of DAA | 12 weeks after the treatment with DAA regimen
  Sustained virological response at 12 week; ie, HCV RNA <15 IU/ ml at 12 weeks after the treatment with DAA regimen.

CONTACTS AND LOCATIONS:
Overall Officials: Qing Xie, MD, Principal Investigator — Director of Department of Infectious Disease, Rui Jin Hospital
Locations (11):
- China (11):
  - Changzhou Third People's Hospital, Changzhou, Jiangsu
  - The Second Hospital of Nanjing, Nanjing, Jiangsu
  - Nanjing Drum Tower Hospital, Nanjing, Jiangsu
  - Jiangsu Province Hospital, Nanjing, Jiangsu
  - The Fifth People's Hospital of Suzhou, Suzhou, Jiangsu
  - Wuxi No. 5 People's Hospital, Wuxi, Jiangsu
  - Rui Jin Hospital Affiliated to Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality
  - Huashan Hospital, Shanghai, Shanghai Municipality
  - Shanghai Public Health Clinical Center, Shanghai, Shanghai Municipality
  - The First Hospital of Jiaxing, Jiaxing, Zhejiang
  - Hwa Mei Hospital, Ningbo, Zhejiang

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lu J, Zhou Y, Lin X, Jiang Y, Tian R, Zhang Y, Wu J, Zhang F, Zhang Y, Wang Y, Bi S. General epidemiological parameters of viral hepatitis A, B, C, and E in six regions of China: a cross-sectional study in 2007. PLoS One. 2009 Dec 24;4(12):e8467. doi: 10.1371/journal.pone.0008467. PMID 20041146
- [Background] Chen YS, Li L, Cui FQ, Xing WG, Wang L, Jia ZY, Zhou MG, Gong XH, Wang FZ, Zheng H, Luo HM, Bi SL, Wang N, Yang WZ, Liang XF. [A sero-epidemiological study on hepatitis C in China]. Zhonghua Liu Xing Bing Xue Za Zhi. 2011 Sep;32(9):888-91. Chinese. PMID 22340876
- [Background] Rao HY, Li H, Chen H, Shang J, Xie Q, Gao ZL, Li J, Sun Y, Jiang J, Wang L, Zhao L, Zhang L, Yang W, Niu J, Gong Z, Gong G, Yang R, Lee MH, Wei L. Real-world treatment patterns and clinical outcomes of HCV treatment-naive patients in China: an interim analysis from the CCgenos study. J Gastroenterol Hepatol. 2017 Jan;32(1):244-252. doi: 10.1111/jgh.13467. PMID 27289083
- [Background] Lu L, Nakano T, He Y, Fu Y, Hagedorn CH, Robertson BH. Hepatitis C virus genotype distribution in China: predominance of closely related subtype 1b isolates and existence of new genotype 6 variants. J Med Virol. 2005 Apr;75(4):538-49. doi: 10.1002/jmv.20307. PMID 15714489
- [Background] Chen Y, Yu C, Yin X, Guo X, Wu S, Hou J. Hepatitis C virus genotypes and subtypes circulating in Mainland China. Emerg Microbes Infect. 2017 Nov 1;6(11):e95. doi: 10.1038/emi.2017.77. PMID 29089588
- [Background] Ogawa E, Furusyo N, Murata M, Hayashi T, Shimizu M, Mukae H, Toyoda K, Hotta T, Uchiumi T, Hayashi J. Impact of HCV kinetics on treatment outcome differs by the type of real-time HCV assay in NS3/4A protease inhibitor-based triple therapy. Antiviral Res. 2016 Feb;126:35-42. doi: 10.1016/j.antiviral.2015.12.001. Epub 2015 Dec 12. PMID 26692214
- [Background] Matthews SJ, Lancaster JW. Telaprevir: a hepatitis C NS3/4A protease inhibitor. Clin Ther. 2012 Sep;34(9):1857-82. doi: 10.1016/j.clinthera.2012.07.011. Epub 2012 Aug 28. PMID 22951253
- [Background] Heo YA, Deeks ED. Sofosbuvir/Velpatasvir/Voxilaprevir: A Review in Chronic Hepatitis C. Drugs. 2018 Apr;78(5):577-587. doi: 10.1007/s40265-018-0895-5. PMID 29546556
- [Background] Feld JJ, Jacobson IM, Hezode C, Asselah T, Ruane PJ, Gruener N, Abergel A, Mangia A, Lai CL, Chan HL, Mazzotta F, Moreno C, Yoshida E, Shafran SD, Towner WJ, Tran TT, McNally J, Osinusi A, Svarovskaia E, Zhu Y, Brainard DM, McHutchison JG, Agarwal K, Zeuzem S; ASTRAL-1 Investigators. Sofosbuvir and Velpatasvir for HCV Genotype 1, 2, 4, 5, and 6 Infection. N Engl J Med. 2015 Dec 31;373(27):2599-607. doi: 10.1056/NEJMoa1512610. Epub 2015 Nov 16. PMID 26571066